CLINICAL TRIAL: NCT00797940
Title: Phase II, Multi-center, Open-Label, Single-Arm Study of Intratumoral Infusion of PRX321 in Subjects With Glioblastoma Multiforme at First Recurrence or Progression
Brief Title: Convection Enhanced Localized Administration of PRX321 With Real-time Imaging for Therapy of Recurrent Glioblastoma (CLARITY-1)
Acronym: CLARITY-1
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No funding for study
Sponsor: Sophiris Bio Corp (Industry)
Responsible Party: Sponsor
Organization: Protox Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRX321-1-05
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Glioblastoma Multiforme
Keywords: GBM; Glioblastoma; Glioblastoma Multiforme; Brain Tumor; Brain Cancer; Glioma
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Up to 42 subjects with first recurrence or progression of GBM
  Interventions: Drug: IL-4PE

INTERVENTIONS:
Drug: IL-4PE — Subjects will receive intratumoral infusion of PRX321 administered via convection-enhanced delivery (CED) at a concentration of 1.5 μg/mL and a total volume of 60 mL over 2 to 7 days.
  Other Names: PRX321

SUMMARY:
A Phase II, multi-center, open-label, single-arm study in up to 42 subjects with first recurrence or progression of GBM at up to 12 sites in Australia, Europe, Israel, and the United States. Subjects will receive intratumoral infusion of PRX321 administered via convection-enhanced delivery (CED) at a concentration of 1.5 μg/mL and a total volume of 60 mL over 2 to 7 days.

Primary Objective:

To evaluate the efficacy (expressed as overall survival at 6 months [OS-6]) of intratumoral infusion of PRX321 in subjects with first recurrence or progression of glioblastoma multiforme (GBM).

Secondary Objectives:

To assess the safety of intratumoral infusion with PRX321 in subjects with recurrent or progressive GBM.

To evaluate objective response rate (ORR), duration of response (DR), overall survival (OS), and progression-free survival (PFS).

Tertiary Objective:

To evaluate the relationship of observed infusate distribution with clinical and radiological responses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects at least 18 years old
* GBM at first recurrence or progression (i.e., disease progressed after any first-line therapy including surgery and radiotherapy as confirmed by MR imaging [MRI]); screening MRIs used to confirm eligibility must be available to the Investigator and the Independent Review Committee (IRC)
* Unilateral, unifocal, and supratentorial tumor, with a maximum diameter of 4 cm (i.e., maximum distance between the borders/edges of enhancing regions) visualized in any arbitrary imaging plane, as assessed by the IRC on MRI taken pre-study 2 weeks prior to catheter placement
* Histological confirmation of GBM (confirmation before primary therapy is acceptable)
* KPS ≥ 70
* If female of childbearing potential, an acceptable method of contraception must be combined with negative pregnancy test before entering the study and must be willing to use contraception for 2 months after treatment with PRX321; male subjects who are non-sterile (i.e., male who has not been sterilized by vasectomy for at least 6 months) must be willing to use a barrier method of contraception for at least 2 months after treatment with PRX321. Acceptable methods of contraception are:

  * intra-uterine contraceptive device without hormone release system: placed at least 4 weeks prior to treatment with PRX321;
  * simultaneous use of male condom and diaphragm + spermicide: starting at least 14 days prior to treatment with PRX321; or
  * simultaneous use of male condom and female condom + spermicide: starting at least 14 days prior to treatment with PRX321
* Able to read, understand, and sign the informed consent document before undergoing any study-specific procedures or have a legal representative willing to do so
* Able and willing to undergo multiple MRI examinations
* Able and willing to comply with all study procedures

Exclusion Criteria:

* A tumor in the brain stem (not including fluid attenuation inversion recovery [FLAIR] changes), an infratentorial tumor, or multifocal satellite tumors
* Tumor with a clinically significant mass effect (> 5 mm midline shift) while on a stable corticosteroid dose
* Subjects with tumors that are completely liquefied (cystic or ring enhancement) in which convection would not be possible
* Tumor with geometric features that make them difficult to adequately cover the tumor volume with infusate by using CED catheters; these tumors include the following:

  * Tumors that appear to wrap around ventricular structures, such that the catheter tips may be positioned within 1.0 cm of a ventricle or such that a large angle (such as an "elbow" or "L- shape") in the tumor shape is present and convection is likely to be compromised;
  * Tumors in which post-surgical enhancement in T1 images in the margins around a resection cavity may be confused with recurring tumor; subjects in whom this enhancement exceeds 5 mm thickness are excluded
* Clinical symptoms that are thought by the Investigator to be caused by uncontrolled increased intracranial pressure, hemorrhage, or edema of the brain
* Inadequate organ function, defined as 1 or more of the following:

  * Hemoglobin < 9.0 g/dL (support with therapeutic erythropoietin products is acceptable);
  * Absolute neutrophil count (ANC) < 1500/mm3 (unsupported by colony stimulating factors);
  * Platelet count < 100,000/mm3 (unsupported by colony stimulating factors);
  * Total bilirubin > 2.0 x upper limit of normal (ULN);
  * Alanine transaminase (ALT) and aspartate transaminase (AST) > 3.0 x ULN;
  * Prothrombin time (PT)/international normalized ratio (INR) > 1.5;
  * Creatinine > 3.0 x ULN;
  * glomerular filtration rate (GFR) < 30 mL/min/1.73 m2;
* Received previous treatment with anti-neoplastic chemotherapeutic agents or craniotomy within 4 weeks before catheter placement
* All subjects who had previously been treated with nitrosoureass must have a 6 to 8 week recovery period from prior toxicity before they can enroll into the study
* Have a known sensitivity or allergy to Gd-DTPA
* Received radiation therapy within 8 weeks prior to catheter placement
* Undergone prior radiosurgery boost (e.g., stereotactic radiosurgery) or other locally targeted therapy other than resection (e.g., Gliadel®, Cotara®) within 3 months of catheter placement
* Received investigational drug therapy for GBM within 4 weeks of catheter placement
* Presence of another type of malignancy within less than 5 years prior to the screening visit, except for adequately treated carcinoma in-situ of the cervix, prostate cancer not actively treated, and basal or squamous cell carcinoma of the skin
* Concurrent or a history of other major disease that could, in the opinion of the Investigator, put the subject at additional risk or interfere with the interpretation of the results of this trial
* Unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's returning for follow-up visits or other unspecified reasons that, in the opinion of the Investigator or Sponsor, make the subject's enrollment incompatible with study objectives
* Life expectancy of less than 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy (expressed as overall survival at 6 months [OS-6]) of intratumoral infusion of PRX321 in subjects with first recurrence or progression of glioblastoma multiforme (GBM) | 6 months

SECONDARY OUTCOMES:
To evaluate objective response rate (ORR), duration of response (DR), overall survival (OS), and progression-free survival (PFS). To assess the safety of intratumoral infusion with PRX321 in subjects with recurrent or progressive GBM. | Up to 24 months